CLINICAL TRIAL: NCT01810887
Title: A Study to Evaluate the Pharmacokinetics and Safety of Oral Single-Dose JNS011 Tablet in Combination With Low-Dose Ritonavir Capsule in Healthy Japanese Adult Males
Brief Title: A Phase 4 Study to Evaluate Pharmacokinetics and Safety of Darunavir Along With Ritonavir in Healthy Male Japanese Participants
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Janssen Pharmaceutical K.K. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR100323; JNS011-JPN-01
Record Dates: First submitted 2013-03-12; First posted 2013-03-14 (Estimated); Last update posted 2013-04-10 (Estimated); Status verified 2013-04

CONDITIONS: Healthy
Keywords: Healthy; Darunavir; JNS011; Ritonavir
MeSH Terms: interventions — Darunavir; Ritonavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ritonavir and darunavir (Experimental): Ritonavir will be administered orally twice daily at a dose of 100 milligram (mg) from Day 1-5. Darunavir ethanolate will be administered as single oral dosing of two tablets of 300 mg on Day 3.
  Interventions: Drug: Darunavir; Drug: Ritonavir

INTERVENTIONS:
Drug: Darunavir — Darunavir ethanolate will be administered as single oral dosing of two tablets of 300 milligram (mg) on Day 3.
  Other Names: JNS011
Drug: Ritonavir — Ritonavir capsule will be administered orally twice daily at a dose of 100 mg for 5 days.
  Other Names: Ritonavir will be administered orally twice daily as 100 mg capsule from Day 1-5.

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetics (explores what the body does to the drug) and safety of darunavir, and will be administered in combination with Ritonavir in healthy adult Japanese male participants.

DETAILED DESCRIPTION:
This is an open-label (all people know the identity of the intervention), single oral-dose and post-marketing study of darunavir administered in combination with low-dose ritonavir in healthy adult Japanese male participants. The total study duration will be approximately of 14 days per participant. The study consists of 3 parts: Screening (that is, 28 days before study commences on Day 1); Treatment (that is, Day 1-5); and Follow-up (that is, up to Day 13). The participants will be hospitalized for 6 nights and 7 days. All the eligible participants will receive Darunavir oral tablet on Day 3 and ritonavir capsule orally twice daily from Day 1-5. Participants will keep upright position until 4 hours after study drug administration. Both the drugs will be administered within 15 minutes after completion of meal. Blood samples will be collected for evaluation of pharmacokinetics at pre-dose and post-dose of study treatment. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Male Participants provided with sufficient explanation of the investigational product, the drugs to be provided and this clinical study prior to the start of participation in the clinical study, and capable of providing voluntary informed consent in writing
* Male Participants with a Body Mass Index (BMI) between 18.5 and 25.0 kilogram per square meter (kg/m^2) at the time of the Screening tests
* Non-smokers or male participants who are capable of abstaining from smoking during the period from the day before the Screening tests until the completion of the post-treatment examinations
* Male Participants consenting to use a medically-approved contraceptive method (such as condoms or the like) during the period from hospital admission until the completion of the post-treatment examinations
* Male Participants showing no clinically significant abnormalities at the time of Screening, on the day prior

Exclusion Criteria:

* Participants suffering or with a history of diseases related to the liver, kidneys, circulatory system, respiratory system, digestive system, neuropsychiatric system, hematopoietic function or endocrine function and who may be inappropriate for participation in this clinical study
* Participants who participated in another clinical study and were treated with another investigational product within 120 days prior to the start of the initial dosing of the provided drugs
* Participants giving 200 milliliter (mL) or more of blood within 30 days prior to the start of the initial dosing of the provided drugs or giving 400 mL or more of blood within 90 days prior to the start of the initial dosing of the provided drugs (such as blood donation), or giving a total of 1200 mL or more of blood within the past year
* Participants with a history of hypersensitivity to sulfonamide drugs, drug allergies or drug hypersensitivity, alcohol, pharmaceutical or drug addiction, or who may be addicted
* Participants with positive results for Human Immunodeficiency Virus antigen or antibodies, Hepatitis C Virus antibodies, Hepatitis B Surface antigen or the serological test for syphilis

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2008-05; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Change in Plasma Darunavir Concentration | 0 hour (pre-dose) and 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 9, 12, 24, 48 and 72 hours post-dose of darunavir on Day 3
  Plasma concentration of Darunavir will be determined by collecting blood samples at the defined time points.
Maximum Plasma Concentration (Cmax) of Darunavir | 0 hour (pre-dose) and 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 9, 12, 24, 48 and 72 hours post-dose of darunavir on Day 3
  The Cmax is the maximum plasma concentration.
Area Under the Plasma Concentration-Time Curve From Time Zero to Infinite Time (AUC [0-infinity]) of Darunavir | 0 hour (pre-dose) and 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 9, 12, 24, 48 and 72 hours post-dose of darunavir on Day 3
  The AUC (0-infinity) is the area under the plasma concentration-time curve from time zero to infinite time, calculated as the sum of AUC(last) and C(last)/lambda(z), wherein AUC(last) is area under the plasma concentration-time curve from time zero to last quantifiable time; and C(last) is the last observed quantifiable concentration; and lambda(z) is elimination rate constant.
Terminal Half-Life(t[1/2]) of Darunavir | 0 hour (pre-dose) and 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 9, 12, 24, 48 and 72 hours post-dose of darunavir on Day 3
  Terminal half-life (t[(1/2]) is defined as 0.693/Lambda(z).
Time to reach maximum concentration (tmax) of Darunavir | 0 hour (pre-dose) and 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 9, 12, 24, 48 and 72 hours post-dose of darunavir on Day 3
  The Tmax is time to reach the maximum plasma concentration.
Area Under the Plasma Concentration-Time Curve From Time Zero to Infinite Time (AUC [0-last]) of Darunavir | 0 hour (pre-dose) and 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 9, 12, 24, 48 and 72 hours post-dose of darunavir on Day 3
  The AUC (0-last) is the area under the plasma concentration-time curve from time zero to last quantifiable time, calculated as the sum of AUC(last) and C(last)/lambda(z), wherein AUC(last) is area under the plasma concentration-time curve from time zero to last quantifiable time; and C(last) is the last observed quantifiable concentration; and lambda(z) is elimination rate constant.
Apparent total body clearance (CL/F) of Darunavir | 0 hour (pre-dose) and 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 9, 12, 24, 48 and 72 hours post-dose of darunavir on Day 3
  Clearance is a quantitative measure of the rate at which a drug substance is removed from the body. The CL/F will be calculated by dividing the dose by AUC (0-infinity)
Apparent volume of distribution at the terminal Phase (Vd[z] /F) of Darunavir | 0 hour (pre-dose) and 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 9, 12, 24, 48 and 72 hours post-dose of darunavir on Day 3
  Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired blood concentration of a drug.The Vd(z)/F will be calculated by dividing CL/F by lambda(z).

SECONDARY OUTCOMES:
Change in Plasma Ritonavir Concentration | 0 hour (pre-dose) on Day 1, 2, 3, 4 and 5
  Plasma concentration of Darunavir will be determined by collecting blood samples at the defined time points.
Maximum Plasma Concentration (Cmax) of Ritonavir | 0 hour (pre-dose) on Day 1, 2, 3, 4 and 5
  The Cmax is the maximum plasma concentration.
Time to reach maximum concentration (tmax) of Ritonavir | 0 hour (pre-dose) on Day 1, 2, 3, 4 and 5
  The Tmax is time to reach the maximum plasma concentration.
Area Under the Plasma Concentration-Time Curve From Time Zero to 12 hours (AUC [0-12]) of Ritonavir | 0 hour (pre-dose) on Day 1, 2, 3, 4 and 5
  The AUC (0-12) is the area under the plasma concentration-time curve from time zero to 12 hours, calculated as the sum of AUC(last) and C(last)/lambda(z), wherein AUC(last) is area under the plasma concentration-time curve from time zero to last quantifiable time; and C(last) is the last observed quantifiable concentration; and lambda(z) is elimination rate constant.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutical K.K., Japan Clinical Trial, Study Director — Janssen Pharmaceutical K.K.
Locations (1):
- Tsukuba, Japan